CLINICAL TRIAL: NCT00352066
Title: A Phase I, Open Label, Controlled, Intra-subject Comparison Study to Investigate the Effect of Co-administration Upon the Pharmacokinetics of Tipranavir (Ritonavir Boosted) and Apricitabine.
Brief Title: Pharmacokinetics of Apricitabine and Tipranavir When Dosed Alone or Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avexa (Industry)
Responsible Party: Susan Cox, Avexa
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AVX-102
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infection
Keywords: Human Immunodeficiency Virus; anti-retroviral therapy; nucleoside analogue; reverse transcriptase; apricitabine; tipranavir; bioequivalence; drug-drug interaction; pharmacokinetics
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — apricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: apricitabine

SUMMARY:
The aim of the study is to see if apricitabine or tipranavir affect the levels of each other in the blood (pharmacokinetic interaction) when they are dosed together.

DETAILED DESCRIPTION:
Apricitabine is a new NRTI in development for treatment of drug resistant HIV. Tipranavir is a recently licensed protease inhibitor for treatment of drug resistant HIV. Tipranavir affects the plasma concentration of some other drugs when they are used together with tipranavir. This study will examine whether the pharmacokinetics of apricitabine are changed when it is dosed together with tipranavir compared to apricitabine alone. Also, the pharmacokinetics of tipranavir will be examined at steady state when it is dosed alone and when it is dosed together with apricitabine. Information on the safety and tolerability of the two drugs when dosed together will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* healthy males 18-40 years old
* non-smokers
* no clinically significant medical history

Exclusion Criteria:

* current or relevant previous medical history of significance
* hepatitis B, hepatitis C, or HIV positive
* current use of prescription or OTC medications
* use of illicit substances or alcohol (>14 drinks/week)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To compare the single dose pharmacokinetics of apricitabine when administered alone and in the presence of steady state concentrations of tipranavir 500 mg administered twice daily in combination with ritonavir 200 mg twice daily. | day 1 and day 10

SECONDARY OUTCOMES:
To compare the steady state pharmacokinetics of tipranavir 500 mg administered twice daily with ritonavir 200mg in the presence and absence of apricitabine. | day 9 and day 10
To evaluate the safety and tolerability of apricitabine administered in combination with tipranavir and ritonavir. | day 10

CONTACTS AND LOCATIONS:
Overall Officials: Susan W Cox, Ph D, Study Director — Avexa
Locations (1):
- Jasper Clinic Inc, Kalamazoo, Michigan, United States